CLINICAL TRIAL: NCT06520163
Title: A Prospective, Multicenter, Randomized Controlled Trial Comparing the Efficacy and Safety of Etoposide, Cytarabine, and PEG-rhG-CSF Combination Therapy vs. Disease-Specific Chemotherapy for Hematopoietic Stem Cell Mobilization in Lymphoma
Brief Title: Comparison Study of EAP and Disease-Specific Chemotherapy Regimens in Hematopoietic Stem Cell Mobilization for Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Affiliated People's Hospital of Ningbo University (Other Government)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Jinhua People's Hospital (Other); The Central Hospital of Lishui City (Other); Shaoxing People's Hospital (Other); Shaoxing Second Hospital (Other); Zhejiang Provincial Tongde Hospital (Other); Taizhou Hospital (Other); Dongyang People's Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Huzhou Central Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Jinhua Municipal Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-059
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Non-Hodgkin's Lymphoma; Hematopoietic Stem Cell Mobilization
Keywords: Non-Hodgkin's Lymphoma; Disease-Specific Chemotherapy; Hematopoietic stem cell mobilization; Etoposide, Cytarabine Combined with PEG-rhG-CSF
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Etoposide; Cytarabine; pegylated granulocyte colony-stimulating factor; Granulocyte Colony-Stimulating Factor; CVAD protocol; EPOCH protocol; Guanosine Diphosphate; 1-(1-glycero)dodeca-1,3,5,7,9-pentaene; Ice

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, two-arm, multicenter, exploratory study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EAP regimen group (Experimental): 66 subjects will be enrolled into the EAP regimen group. EAP regimen is the etoposide, cytarabine, and PEG-rhG-CSF combination therapy.
  Interventions: Drug: Etoposide; Drug: Cytarabine; Drug: PEG-rhG-CSF; Drug: G-CSF
- Disease-specific chemotherapy mobilization regimens group (Active Comparator): 33 subjects will be enrolled into the disease-specific chemotherapy mobilization regimens group. The disease-specific chemotherapy mobilization regimens include but not limited to: CHOP, Hyper-CVAD, ID-MTX+Ara-C.
  Interventions: Combination Product: CHOP; Combination Product: Hyper-CVAD; Combination Product: ID-MTX + Ara-C; Combination Product: DA-EPOCH; Combination Product: GDP; Combination Product: GDPE; Combination Product: ICE; Combination Product: DICE; Drug: G-CSF

INTERVENTIONS:
Drug: Etoposide — Day 1~Day 2: 75mg/m^2
  Other Names: VP-16
  Arms: EAP regimen group
Drug: Cytarabine — Day 1~Day 2: 200g/m^2, q12h
  Other Names: Ara-C
  Arms: EAP regimen group
Drug: PEG-rhG-CSF — Day 6: 6mg
  Arms: EAP regimen group
Drug: G-CSF — Starting from the 9th day, if the white blood cell count is less than 20,000/μL, administer G-CSF at a dose of 5μg/kg by subcutaneous injection until the collection is completed.
  Arms: EAP regimen group
Combination Product: CHOP — [Cyclophosphamide (Cy) + Doxorubicin (ADM) + Vincristine (VDS) + Prednisone (Pred) ]± Rituximab (R)
  Arms: Disease-specific chemotherapy mobilization regimens group
Combination Product: Hyper-CVAD — [Cyclophosphamide + Doxorubicin + Vincristine + Dexamethasone (DXM)] ± Rituximab
  Arms: Disease-specific chemotherapy mobilization regimens group
Combination Product: ID-MTX + Ara-C — [High-Dose Methotrexate (MTX) + Cytarabine] ± Rituximab
  Arms: Disease-specific chemotherapy mobilization regimens group
Combination Product: DA-EPOCH — [Etoposide + Doxorubicin + Vincristine + Cyclophosphamide + Prednisone] ± Rituximab
  Arms: Disease-specific chemotherapy mobilization regimens group
Combination Product: GDP — [Gemcitabine (G) + Cisplatin (P) + Dexamethasone (DXM)] ± Rituximab
  Arms: Disease-specific chemotherapy mobilization regimens group
Combination Product: GDPE — [Gemcitabine + Cisplatin + Dexamethasone + Etoposide] ± Rituximab
  Arms: Disease-specific chemotherapy mobilization regimens group
Combination Product: ICE — [Etoposide + Ifosfamide (IFO) + Carboplatin] ± Rituximab
  Arms: Disease-specific chemotherapy mobilization regimens group
Combination Product: DICE — [Dexamethasone + Ifosfamide + Ifosfamide + Etoposide] ± Rituximab
  Arms: Disease-specific chemotherapy mobilization regimens group
Drug: G-CSF — From Day 6, administer G-CSF at a dose of 5μg/kg by subcutaneous injection until the collection is completed.
  Arms: Disease-specific chemotherapy mobilization regimens group

SUMMARY:
This study utilizes a prospective, multicenter, randomized two-arm design to evaluate the efficacy and safety of the etoposide, cytarabine, and pegylated recombinant human granulocyte colony-stimulating factor (PEG-rhG-CSF) combination therapy (EAP regimen) in mobilizing hematopoietic stem cells in patients with non-Hodgkin's lymphoma (NHL). A total of 99 NHL patients will be enrolled as research subjects and will be randomly allocated in a 2:1 ratio to compare the EAP regimen versus disease-specific chemotherapy mobilization regimen. The primary endpoint is the proportion of patients achieving the ideal collection value after a single collection (CD34+ cells ≥5×10^6/kg).

DETAILED DESCRIPTION:
Based on strict inclusion and exclusion criteria, a total of 99 non-Hodgkin's lymphoma patients from 16 hospitals will be selected. Eligible subjects will be randomly assigned in a 2:1 ratio to either the experimental group or the control group. The experimental group will receive the EAP regimen, which combines etoposide, cytarabine, and pegylated recombinant human granulocyte colony-stimulating factor (PEG-rhG-CSF), while the control group will receive disease-specific chemotherapy mobilization regimens, such as the CHOP and Hyper-CVAD. Subsequently, the number of CD34+ cells will be monitored. The study will evaluate the proportion of patients achieving the ideal collection value after a single collection (CD34+ cells ≥5×106/kg); the proportion of patients achieving the target collection value cumulatively; the total amount of CD34+ cells collected and the average number of collections; hematological and non-hematological adverse reactions; and the proportion of patients receiving plerixafor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with non-Hodgkin's lymphoma before enrollment.
* Indication for autologous stem cell transplantation (ASCT).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0~1.
* Achieved complete remission after multiple courses of chemotherapy.
* Life expectancy ≥ 3 months.
* Subjects must be able to understand the protocol and sign the informed consent.

Exclusion Criteria:

* Cardiac function class II or higher or cardiac ejection fraction < 40%.
* Serum direct bilirubin (DBIL) more than twice of the upper limit of normal (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) more than three times the upper limit of normal (ULN).
* Serum creatinine clearance rate ≤ 50%.
* Patients with active infection.
* History of prior hematopoietic stem cell mobilization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
% of patients achieving the collection of ≥5×10^6 CD34+ cells/kg | 1 month
  Proportion of patients who achieve the ideal collection value (CD34+ cells ≥5×10^6/kg) after a single collection.

SECONDARY OUTCOMES:
% of patients achieving the collection of ≥2×10^6 CD34+ cells/kg | 1 month
  To observe and compare the proportion of patients who cumulatively achieve the target collection value (CD34+ cells ≥ 2×10^6/kg) between the EAP regimen and the disease-specific chemotherapy regimen; the proportion of patients who achieve the ideal collection value.
CD34+ cells and the average number of collections | 1 month
  To observe and compare the total cumulative collection of CD34+ cells and the average number of collections between the EAP regimen and the disease-specific chemotherapy regimen.
Adverse Rvents (AEs) | 1 month
  To observe and compare the hematological and non-hematological adverse reactions between the EAP regimen and the disease-specific chemotherapy regimen.
% of patients who use Plerixafor | 1 month
  To observe and compare the proportion of patients who receive plerixafor added to the EAP regimen and the disease-specific chemotherapy regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Peipei Ye, Principal Investigator — The Affiliated People's Hospital of Ningbo University
Locations (17):
- China (17):
  - Dongyang People's Hospital, Dongyang, Zhejiang
  - The Affiliated Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Tongde Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Huzhou central hospital, Huzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Jinhua People's Hospital, Jinhua, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - The Affiliated People's Hospital of Ningbo University, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Shaoxing Second Hospital, Shaoxing, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou